CLINICAL TRIAL: NCT03710967
Title: Bilateral vs. Unilateral Transcranial Magnetic Stimulation of the Primary Motor Cortex to Treat Chronic Orofacial Pain: a Pilot Study With a Randomized Controlled Design
Brief Title: Bilateral TMS vs. Unilateral TMS
Acronym: biTMSvsuniTMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL62849.091.17
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-06

CONDITIONS: Neuropathic Pain; Orofacial Pain; Trigeminal Neuropathy
MeSH Terms: conditions — Neuralgia; Facial Pain; Trigeminal Nerve Diseases | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: single-blinded, randomized controlled cross-over design trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral TMS (Experimental)
  Interventions: Device: Transcranial magnetic stimulation
- Unilateral TMS (Active Comparator)
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Transcranial magnetic stimulation of the primary motor cortex

SUMMARY:
Rationale: In 2016, Henssen et al. discuss that orofacial pain may be conducted in a bilateral fashion, inducing activation of both thalami [1]. For this reason, bilateral stimulation of the motor cortex is thought to induce a stronger analgesic effect compared to unilateral motor cortex stimulation by transcranial magnetic stimulation.

Objective: To investigate the superiority of bilateral transcranial magnetic stimulation (TMS) over unilateral TMS of the motor cortex Study design: Double-blind, randomized controlled trial Study population: Patients that suffer from chronic orofacial pain and have not been treated (yet) with any form of neuromodulation.

Intervention (if applicable): One group receives bilateral TMS whereas the other group receives unilateral TMS for one month. After one month, the groups switch treatment protocol.

Main study parameters/endpoints: Modification in intensity of pain as measured using the VAS, the influence the relief of pain with regard to quality of life and daily activities using the McGill Pain Questionnaire.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Time investment of patients.

DETAILED DESCRIPTION:
For this study, we aim to include 12 patients with intractable, chronic orofacial pain of peripheral origin with a baseline VAS of at least 5 (0= no pain, 10= worst possible pain). The investigator (Dylan Henssen) contacts the pain nurse, neurosurgeons and pain physicians to ask them to seek contact with their patients to inform them about this research. Afterwards, if the patients wish to learn more or wish to participate, they receive an information package, including an information letter and an informed consent form. When the patient agrees to be included they receive four McGill Pain questionnaires which must be filled in weekly. After these four weeks, the patient is invited to the outpatient clinic to meet with the investigator. During this consultation, the patient talks about the pain he/she experiences, submits the four filled-in questionnaires and receives further information about the research. After the consultation, all patients are randomized in double-blinded fashion.

At the next meeting at the Donders Institute at Nijmegen, the patient takes place in a relaxing chair. A second, independent researcher will install the transcranial magnetic stimulation (TMS) coils, one on each side of the patient. The coils are positioned in such a fashion that both the coils can stimulate the primary motor cortex. Then the independent researcher starts the stimulation protocol. In the first session, the patient either receives unilateral or bilateral stimulation. After this session, the patient fills in a new McGill Pain questionnaire in order to measure the pain sensation after the first session of TMS. Then the patient goes home for one month. At home, another 4 McGill Pain Questionnaires are asked to fill in. After this, the patient returns to the Donders Institute to take place in the relaxing chair in order to be treated in the second session. Again, the patient either receives unilateral or bilateral stimulation, depending on what was received during the first session. Again, the patients are asked to fill in 4 new McGill Pain questionnaires, one per week (See figure 1).

At the end of this session, the patient is invited to meet with the investigator or independent researcher once more to talk about their experiences and pain relief during the research. This interview takes place at Radboudumc and is audio recorded.

All the McGill Pain questionnaires are analyzed by the researcher (Dylan Henssen) using SPSS. Afterwards, the independent researcher discloses which patient received uni- or bilateral in which order. The audio recorded interviews are transcribed verbatim and analyzed using Atlas.tii.

ELIGIBILITY:
Inclusion Criteria:

1. Suffering from painful trigeminal neuropathy according to the International Classification of Headache Disorder (ICHD), 3rd beta version;
2. Mean pain-intensity scores at baseline needed to be greater than 50mm as measured by the visual analogue scale (VAS);
3. Aged between 18-80 years old;
4. Non-pregnant, non-lactating and not planned to become pregnant during the study;
5. Capable of completing headache pain self-assessments;
6. Agrees not to change any medication or dosages in relation to the painful trigeminal neuropathy during the study

Exclusion Criteria:

Patients were excluded from this study when they suffered from other neurological diseases (i.e., multiple sclerosis or epilepsy) or other chronic pain conditions or had a history of intracranial aneurysm, intracranial hemorrhage, brain tumor, or significant head trauma. Other exclusion criteria concerned patients having a pacemaker, intracardial device, neuromodulation device or other forms of metal implants in the craniocervical region. Finally, only patients who did not undergo any form of TMS prior to this experiment were included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 8 weeks
  Visual analogue scale

SECONDARY OUTCOMES:
Medication intake | 8 weeks
  Medication quantification scale
Quality of life | 8 weeks
  McGill Pain Questionnaire: Quality of life index
Pain descriptor | 8 weeks
  McGill Pain Questionnaire: Pain descriptors

OTHER OUTCOMES:
Patient global improvement scale | 8 weeks
  PGIC
Qualitative assessment | 8 weeks
  Face-to-face interviews

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Henssen, MD, Principal Investigator — RadboudUniversity
Locations (1):
- Radboud University, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided